CLINICAL TRIAL: NCT00281112
Title: Center for Reducing Asthma Disparities - Howard/Hopkins Centers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1196; U01HL072433-04 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To evaluate asthma morbidity in low-income, African-American children and adults with asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition affecting over 14 million Americans, but the prevalence rates are higher in certain populations (e.g. 10 percent in inner-cities and 30 percent among the homeless vs. 5 percent in a general population of whites). African Americans and Hispanics from the Northeast are twice as likely to die from asthma as whites. African Americans are four times as likely to be hospitalized for asthma and are five times more likely than whites to seek care for asthma at an emergency department. Reasons for these higher rates are not certain, and most likely result from an interaction of risk factors such as environmental exposures, genetic predisposition, access to appropriate medical care, socioeconomic status, and cultural health practices. The National Heart, Lung, and Blood Institute supports a variety of activities to address the pressing public health problems posed by asthma. However, progress in reducing disparities has been disappointingly slow. Separate, independent research projects have generated important clues for understanding the nature and scope of the problem. A more coordinated, interdisciplinary and comprehensive approach to research is needed to take advantage of these clues, move the science further and faster, and increase our capacity to improve health outcomes among minority and economically disadvantaged populations. Cooperative centers of research that foster partnerships among minority medical centers, research intensive institutions, and the communities in which asthma patients live will promote such advancement.

The Request for Applications for the Centers for Reducing Asthma Disparities was released in October, 2001. The objective of the program is to promote partnerships (called Centers) between a minority serving institution (MSI) that may not have a strong research program and a research intensive institution (RII) that has a track record of NIH-supported research and patient care. The purpose of the partnership is to conduct collaborative research on asthma disparities (i.e. greater prevalence of asthma, higher rates of morbidity due to asthma, and lesser access or use of quality medical care among minorities and poor).

DESIGN NARRATIVE:

The center has four research projects designed to collaboratively investigate factors associated with the disproportionate burden of asthma experienced by inner-city, African-American children and adults. This includes studies that will evaluate both the underlying genetic factors that may contribute to the observed excess risk in African-American communities, as well as studies of provider-patient communication designed to assess intervention strategies for remediating this risk. In addition, an essential goal of the Howard/Hopkins Center for Reducing Asthma Disparities will be to create a culturally sensitive training environment that is truly reciprocal, and designed to both enrich and enhance the research potential and asthma management capabilities of both participating institutions.

Research project 1 will create and validate a culturally sensitive and simple to administer Asthma Communication Instrument for use in describing asthma symptoms. Research project 2 will develop a tripartite communication mechanism between the patient, the patient care provider, and an asthma counselor. Research project 3 deals with the genetics of cockroach allergy. Research project 4 will develop a complementary mouse model to address the role of the genetics of cockroach sensitization as it pertains to asthma disparities.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Floyd Malveaux — Howard University; Cynthia Rand — Johns Hopkins University